CLINICAL TRIAL: NCT07374185
Title: A New Regenerative Medicine Protocol Using Autologous Bone Marrow Mononuclear Cells With Growth Factors to Treat Liver Cirrhosis
Brief Title: Using Autologous Bone Marrow Cells With Wharton Gel Exosomes to Stimulate Hepatic Cell Repair in Liver Cirrhosis
Acronym: bone marrow
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Global Stem Cell Center, Baghdad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ifaa-stem protocol
Record Dates: First submitted 2025-11-28; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: 10 cases liver cirrhosis regardless of the stage to be treated with autologous cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- active treatment cellular product arm (Active Comparator): autologous bone marrow aspiration is done under sedation with the addition of Wharton gel 2 cc exosomes then given intravenously after using 170 micron filter.
  Interventions: Procedure: Autologous Bone Marrow Aspirate Concentrate

INTERVENTIONS:
Procedure: Autologous Bone Marrow Aspirate Concentrate — using autologous bone marrow aspirated from iliac crest ,centrifuged and then injected intravenously

SUMMARY:
the study includes patients with liver cirrhosis irrespective of the stage excluding people with active tumor or other major health issue endangering life, the protocol includes the use of autologous bone marrow derived mononuclear cells harvested from the same patient under local anesthesia ,followed by cell concentration and viability testing , then final product is combined with small volume of 2 cc of Wharton gel exosomes 20 billion per to be administered intravenously.

DETAILED DESCRIPTION:
Mesenchymal stem cell therapy is one option that can help in improving liver functions if given parenteral, those mesenchymal stem cells can be harvested from different sources ,regarding this trial investigators use bone marrow derived mononuclear cells taken from posterior crest of iliac bone of the same patient, the bone marrow volume taken is around 50 cubic milliliter to be followed by filtration to get rid of bone fragments then Wharton gel exosomes are added in 2 cc volume and total 20 billion particles ,the product is administered intravenously .

ELIGIBILITY:
Inclusion Criteria: any patient with liver cirrhosis , less than 80 years of age -

Exclusion Criteria:

1. active malignancy.
2. severe sepsis.
3. pregnancy. -

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
child-Pugh score for liver cirrhosis | 12 weeks up to 12 months
  The Child-Pugh score is a clinical tool used to assess the severity and prognosis of chronic liver disease, especially cirrhosis, by evaluating five key factors: total bilirubin, albumin, INR (prothrombin time), ascites, and hepatic encephalopathy, with each getting 1-3 points (1=best, 3=worst). Summing these points categorizes patients into Class A (5-6 points, well-compensated), B (7-9 points, moderately impaired), or C (10-15 points, severe dysfunction), helping guide treatment, predict surgical risk, and manage liver transplant needs. A is minimum and C maximum
child-Pugh score of 3 stages depends on bilirubin level, serum albumin ,prothrombin time ,ascites ,encephalopathy | 12 months
  measurement of prothrombin time, albumin, serum bilirubin level and assess ascites and hepatic encephalopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Private Hospital Alrabee Street, Baghdad, Iraq, Iraq

IPD SHARING:
Plan to Share IPD: No